CLINICAL TRIAL: NCT00762307
Title: A Prospective, Multi-Center Clinical Study of Non-Invasive Cooling of Subcutaneous Fat
Brief Title: Non-invasive Cooling of Subcutaneous Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JM07001
Record Dates: First submitted 2008-09-27; First posted 2008-09-30 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2020-09

CONDITIONS: Fat Disorder
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Treatment Group 1 (Experimental): Cooling Intensity Factor = 33 Duration = 60 minutes
  Interventions: Device: Zeltiq Dermal Cooling Device
- Treatment Group 2 (Experimental): Cooling Intensity Factor = 37 Duration = 30 minutes
  Interventions: Device: Zeltiq Dermal Cooling Device
- Treatment Group 3 (Experimental): Cooling Intensity Factor = 37 Duration = 45 minutes
  Interventions: Device: Zeltiq Dermal Cooling Device
- Treatment Group 4 (Experimental): Cooling Intensity Factor = 42 Cooling Duration = 30 minutes
  Interventions: Device: Zeltiq Dermal Cooling Device

INTERVENTIONS:
Device: Zeltiq Dermal Cooling Device — Noninvasive cooling is applied to the treatment area with a defined cooling rate and duration.

SUMMARY:
The purpose of this study is to evaluate a non-invasive cooling device to determine if cold exposure will consistently result in a reduction of subcutaneous fat.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a non-invasive cooling device to determine if cold exposure will consistently result in a reduction of subcutaneous fat using the Zeltiq Dermal Cooling device.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 18 years of age.
2. Subject has clearly visible fat on the flanks, thighs, abdomen, or back.
3. Subject has not had weight change fluctuations exceeding 10 pounds in the preceding month.
4. Subject has read and signed a written informed consent form.

Exclusion Criteria:

1. Subject has had liposuction, or another surgical procedure(s) or mesotherapy in area of intended treatment within the past 2 years.
2. Subject has a known history of subcutaneous injections into the area of intended treatment (e.g., cortisone) within the past 6 months.
3. Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
4. Subject is taking diet pills within the past 6 months.
5. Subject is unable or unwilling to comply with the study requirements.
6. Subject has any dermatological conditions or scars within the location of the test sites that may interfere with the treatment or evaluation.
7. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
8. Patient is pregnant or intending to become pregnant in the next 9 months.
9. Patient is lactating or has been lactating in the past 9 months.
10. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect response or participation in this clinical study, or would pose an unacceptable risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Jiang, Study Chair — Zeltiq Aesthetics
Locations (4):
- United States (4):
  - Investigational Site, Dublin, California
  - Investigational Site, Fremont, California
  - Investigational Site, Pleasanton, California
  - Investigational Site, San Ramon, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4
Started | 28 | 11 | 11 | 10
Completed | 26 | 11 | 11 | 9
Not Completed | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated with CIF 33 for 60 minutes.
Groups:
- Treatment Group 1: Subjects in Treatment Group 1 were treated using a Cooling Intensity Factor (CIF) of 33 for 60 minutes.
- Treatment Group 2: Subjects in Treatment Group 2 were treated using CIF 37 for 30 minutes.
- Treatment Group 3: Subjects in Treatment Group 3 were treated using CIF 37 for 45 minutes.
- Treatment Group 4: Subjects in Treatment Group 4 were treated using CIF 42 for 30 minutes.
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Total
Number analyzed (Participants) | 28 | 11 | 11 | 10 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 11 | 11 | 9 | 58
  >=65 years | 1 | 0 | 0 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 41 [23 to 65] | 44 [26 to 56] | 44 [28 to 55] | 49 [26 to 65] | 44 [23 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 5 | 5 | 19
  Male | 27 | 3 | 6 | 5 | 41
Region of Enrollment [Number; unit: participants]
  United States | 28 | 11 | 11 | 10 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Fat Layer Thickness of the Treated Flank
Description: The change in fat layer thickness as demonstrated by measurement of fat layer layer thickness using ultrasound images taken in the treated area and on the contralateral flank (control) at baseline and at the 6 month follow-up. Data collected on the untreated side and the treated side will be combined to determine the normalized change in fat layer thickness for each subject. The mean percent fat layer reduction across all treatment groups will be presented, as well as for each treatment group.
Time Frame: Baseline and 6 months
Population: The population includes only subjects with evaluable ultrasound data ( >3 valid images at 6 month follow up visit). Group 1 exclusions: 2 Lost To Follow Up and 6 not evaluable; Group 2 exclusions: 1 not evaluable; Group 3 exclusions: 3 not evaluable; Group 4 exclusions: 1 not evaluable and 1 withdrawn from study by Investigator.
Measure: Mean (Standard Error); unit: percent fat layer change
Groups:
- All Groups: All subjects treated in Groups 1, 2, 3 and 4 are combined for this analysis.
- Group 1: CIF 33 for 60 minutes
- Group 2: CIF 37 30 minute duration
- Group 3: CIF 37 duration 45 minutes
- Group 4: CIF 42 30 duration 30 minutes
Arm/Group | All Groups | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 46 | 20 | 10 | 8 | 8
percent fat layer change | -18.7 (1.9) | -22.6 (3.4) | -17.8 (3.6) | -17.5 (2.3) | -11.1 (3.8)
Statistical Analysis 1: Comparison: All Groups; Test type: Other; Mean Difference (Net) = 18.7, 95% CI 2-sided [14.9 to 22.4], Standard Error of Mean 1.9

2. Primary Outcome: Percentage of Subjects Expressing Satisfaction With the Procedure
Description: Subject satisfaction as determined by the completion of a questionnaire at the 6 month follow-up visit, and, as requested, any other follow-up visits.
Time Frame: 6 months post-treatment follow-up visit
Population: 56 subjects completed the questionnaire; 2 subjects were LTFU, 1 subject failed to complete the questionnaire and 1 subject was withdrawn from the study by the Investigator. Four (4) subjects did not respond to one question on the questionnaire; 1 subject did not respond to another question on the questionnaire.
Measure: Mean (Standard Deviation); unit: percent positive responses
Groups:
- Overall Study Population: All subjects treated in Treatment Groups 1,2,3 and 4 are in the Overall Study Population
- Treatment Group 1: Cooling Intensity Factor= 33 Duration of Cooling = 60 minutes
- Treatment Group 2: Cooling Intensity Factor = 37 Cooling Duration = 30 minutes
- Treatment Group 3: Cooling Intensity Factor = 37 Cooling Duration = 45 minutes
Arm/Group | Overall Study Population | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4
Number analyzed (Participants) | 56 | 25 | 11 | 11 | 9
percent positive responses
  Overall satisfaction with treatment experience | 82.1 (5.1) | 84 (7.3) | 81.8 (11.6) | 90.9 (8.7) | 66.7 (15.7)
  Agree there is a change to the treated area: number analyzed (Participants) | 55 | 25 | 11 | 10 | 9
  Agree there is a change to the treated area | 76.3 (5.7) | 84 (7.3) | 54.5 (15.0) | 100 (0) | 55.6 (16.6)
  Agree change to treated area was improvement: number analyzed (Participants) | 52 | 21 | 11 | 11 | 9
  Agree change to treated area was improvement | 78.9 (5.7) | 95.2 (4.7) | 63.6 (14.5) | 81.8 (11.6) | 55.6 (16.6)
  Expectations were met or exceeded | 73.2 (5.9) | 72 (9.0) | 78.6 (12.4) | 81.8 (11.6) | 66.7 (15.7)
  Discomfort was no greater than expected | 98.2 (1.8) | 100 (0) | 90.9 (8.7) | 100 (0) | 100 (0)

3. Primary Outcome: Percentage of Correctly Identified Pre-treatment Photographs
Description: Change in the treated vs. untreated areas will be assessed for changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the control and treated flanks. Reviewers will be practicing dermatologists. All reviewers will be blinded to post-treatment vs. baseline and/or untreated flank. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form.Criteria for evaluable photos for the purposes of the independent review: subject completed treatment regimen; subject has complete set of baseline photos; subject has a complete set of post-treatment photos; photos were taken using Zeltiq standard procedure. Results reflect the percentage of correctly identified images.
Time Frame: Baseline and 6 months
Population: The analysis population included subjects who had evaluable photos from baseline and the 6 month final follow-up visit. Subjects who did not maintain their weight per protocol requirements were excluded from analysis.
Measure: Mean (Standard Error); unit: percent correctly identified images
Groups:
- All Groups: Treatment Groups 1, 2, 3 and 4 were combined for this analysis.
Arm/Group | All Groups | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4
Number analyzed (Participants) | 31 | 11 | 8 | 6 | 6
percent correctly identified images | 91.9 (5.2) | 90.5 (7.6) | 100 (0) | 100 (0) | 83.3 (15.2)
Statistical Analysis 1: Comparison: All Groups; Test type: Other; sucess percentage = 91.9, Standard Error of Mean 5.2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment though the 6 month follow-up visit, a time period of approximately 8 months.
Groups:
- Treatment Group 1: Subjects from Group 1 were treated using a CIF of 33 for 60 minutes in duration.
- Treatment Group 2: Subjects from Group 2 were treated using a CIF of 37 for 30 minutes in duration.
- Treatment Group 3: Subjects in Treatment Group 3 were treated using a CIF of 37 for 45 minutes in duration.
- Treatment Group 4: Subjects in Treatment Group 4 were treated using a CIF of 42 for 30 minutes in duration.
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/11 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/11 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 1/28 | 1/11 | 1/11 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group 1 (N=28) | Treatment Group 2 (N=11) | Treatment Group 3 (N=11) | Treatment Group 4 (N=10)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasm (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No